CLINICAL TRIAL: NCT00190554
Title: A Randomized Controlled Trial of Chemotherapy With 5FU and Cisplatin Before and After Surgery for Stage II,III Squamous Cell Carcinoma of the Thoracic Esophagus:JCOG9907
Brief Title: A Trial of Chemotherapy Before and After Surgery for Stage II,III Esophageal Squamous Cell Carcinoma
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Japan Clinical Oncology Group (Other)
Collaborators: Ministry of Health, Labour and Welfare, Japan (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JCOG9907; C000000223
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Esophageal Neoplasms; Carcinoma, Squamous Cell
Keywords: esophageal cancer; squamous cell carcinoma; esophagectomy; neoadjuvant chemotherapy; esophageal squamous cell carcinoma
MeSH Terms: conditions — Esophageal Neoplasms; Carcinoma, Squamous Cell; Esophageal Squamous Cell Carcinoma | interventions — Fluorouracil; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Surgery +(Cisplatin 80 mg/㎡+5FU 800mg/㎡×5days)×2
Drug: (Cisplatin 80 mg/㎡+5FU 800mg/㎡×5days)×2＋Surgery

SUMMARY:
To determine whether chemotherapy before surgery makes better outcome than chemotherapy after surgery in patients with esophageal squamous cell carcinoma

DETAILED DESCRIPTION:
The previous study JCOG9204 showed that postoperative adjuvant chemotherapy with cisplatin and fluorouracil has a detectable preventive effect on relapse in patients with esophageal squamous cell carcinoma compared with surgery alone.(J Clin Oncol 2003;21:4592-4596) Therefore the standard treatment for stage II and III esophageal cancer is adjuvant chemotherapy after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. histologically proven squamous cell carcinoma of the thoracic esophagus
2. pathologic stages IIa, IIb, III except T4
3. an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
4. no previous history of chemotherapy nor radiotherapy
5. an essentially normal clinical laboratory profile (white blood cell count or WBC, >=4,000 /mm3; hemoglobin or Hb, >=10g/dl; platelet count or Plt, >=100,000 /mm3; total serum bilirubin<=1.2 mg/dl; aspartate aminotransaminase or AST and alanine aminotransaminase or ALT no higher than twice normal; creatinine or CRTN, <=1.2 mg/dl; creatinine clearance or CCr, >=60 ml/minute; and arterial oxygen tension or PaO2, >=65 torr
6. oral or written informed consent obtained before randomization

Exclusion Criteria:

1. severe heart diseases
2. uncontrollable hyper tension or diabetes mellitus
3. severe pulmonary dysfunction
4. HBs positive
5. active bacterial infection
6. synchronous or metachronous (within 5 years) malignancy
7. pregnant female
8. psychiatric medication

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330
Dates: Start 2000-05; Primary Completion 2004-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Disease free survival | year

SECONDARY OUTCOMES:
Overall survival | year
Toxicity of chemotherapy | year
Operative morbidity | year

CONTACTS AND LOCATIONS:
Overall Officials: Nobutoshi Ando, M.D., Study Chair — Tokyo Dental College Ichikawa General Hospital
Locations (24):
- Japan (24):
  - Aichi Cancer Center Hospital, Nagoya,Chikusa-ku,Kanokoden,1-1, Aichi-ken
  - Chiba University, Graduate School of Medicine, Chiba,Chuo-ku,Inohana,1-8-1, Chiba
  - Tokyo Dental College Ichikawa General Hospital, Ichikawashi,Sugano,5-11-13, Chiba
  - National Cancer Center Hospital East, Kashiwa,Kashiwanoha,6-5-1, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama,Horinouchi,13, Ehime
  - Kurume University School of Medicine, Kurume,Asahi-machi,67, Fukuoka
  - Hiroshima City Asa Hospital, Hiroshima,Asakitaku,KabeminamiHiroshima,2-1-1, Hiroshima
  - Iwate Medical University, Morioka,Uchimaru,19-1, Iwate
  - Tokai University School of Medicine, Isehara,Shimokasuya,143, Kanagawa
  - Kanagawa Cancer Center, Yokohama,Asahi-ku,Nakao,1-1-2, Kanagawa
  - Kyoto University Hospital, Kyoto,Sakyo-ku,Syogoinkawara,54, Kyoto
  - Niigata University Medical and Dental Hospital, Niigata,Asahimachi-dori,1-754, Niigata
  - Niigata Cancer Center Hospital, Niigata,Kawagishi-cho,2-15-3, Niigata
  - Osaka National Hospital, Osaka,Chuo-ku,Hoenzaka,2-1-14, Osaka
  - Osaka Medical Center for Cancer and Cardiovascular Diseases, Osaka,Higashinari-ku,Nakamichi,1-3-3, Osaka
  - Sizuoka Cancer Center, Sunto-gun,Nagaizumi-cho,Shimonagakubo,1007, Shizuoka
  - Tochigi Cancer Center, Utsunomiya,Yohnan,4-9-13, Tochigi
  - Juntendo University School of Medicine, Bunkyo-ku,Hongo,3-1-3, Tokyo
  - Tokyo Medical and Dental University Hospital, Bunkyo-ku,Yushima,1-5-45, Tokyo
  - National Cancer Center Hospital, Chuo-ku,Tsukiji,5-1-1, Tokyo
  - National Hospital Organization Tokyo Medical Center, Meguro-ku,Higashigaoka,2-5-1, Tokyo
  - Toranomon Hospital, Minato-ku,Toranomon,2-2-2, Tokyo
  - Tokyo Women's Medical University, Shinjuku-ku,Kawada-cho,8-1, Tokyo
  - Keio University Hospital, Shinjuku-ku,Shinanomachi,35, Tokyo

REFERENCES:
- [Derived] Hirao M, Ando N, Tsujinaka T, Udagawa H, Yano M, Yamana H, Nagai K, Mizusawa J, Nakamura K; Japan Esophageal Oncology Group/Japan Clinical Oncology Group. Influence of preoperative chemotherapy for advanced thoracic oesophageal squamous cell carcinoma on perioperative complications. Br J Surg. 2011 Dec;98(12):1735-41. doi: 10.1002/bjs.7683. Epub 2011 Sep 14. PMID 21918956
- See also: Related Info — http://www.jcog.jp/